CLINICAL TRIAL: NCT05261737
Title: Effectiveness of Steroid Injection in Treating Pain in De Quervain Tenosynovitis
Brief Title: Steroid Injection in De Quervain Tenosynovitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/00787
Record Dates: First submitted 2022-02-14; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: De Quervain Disease
MeSH Terms: conditions — De Quervain Disease | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Corticosteroid Injection — Steroid injection effectiveness will be determined by relief of pain scored by patient using Visual Analogue Scale (VAS). Data will be collected during clinic visit and contacting patients in a determined protocol for the following 6 weeks after steroid injection.After approval of the study, data will collected from participants over a period of 6 weeks follow up; the whole study will be conducted over a total of 2 years.Since the study will not conduct any further test to participants and follow up regimen will only state pain related to the specific condition (De Quervain tenosynovitis) and quick-DASH score, it will not result in any anticipated/unanticipated incidental findings, therefore participants will not be recontacted.

SUMMARY:
This study is carried out to find out the degree of pain relief achieved with standard treatment as steroid injection as well as its time to onset. It will recruit 50 subjects over a period of 18 months.

DETAILED DESCRIPTION:
The aim of the study is determine how effective these injections are and when will the patient start feeling relief of his/her symptoms.The aim of the study is not to change the current practice, but provide hand surgeons enough data to clarify their patients the expected outcomes and onset timing of the treatment performed.

ELIGIBILITY:
Inclusion Criteria:

* >21 years old

Exclusion Criteria:

* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants of the study will be selected by attending physician in Hand and Reconstructive Microsurgery outpatient clinic.
  Estimated sample size is 50 patients.Statistical power calculation (error type II) is 0.8The Kaplan-Meier product-limit method will be used to estimate the rates of freedom from recurrence of symptoms. Confidence intervals for Kaplan-Meier survivorship functions will be based on Greenwood's variance estimated. A multivariable Cox proportional hazards regression model is planned to identify independent predictors of outcome.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-03-14 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Determine efficacy of steroid injection | 7 days
  a single steroid injection over first dorsal compartment for patients diagnosed with de Quervain tenosynovitis will make effect within 7 days from injection, relieving pain to less or equal than 1 in Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Renita Sirisena, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore